CLINICAL TRIAL: NCT02687581
Title: Efficacy of Intermittent Occlusion Therapy Glasses for Amblyopia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment is challenging and study materials were not produced any more.
Sponsor: Salus University (Other)
Collaborators: Indiana University (Other)
Responsible Party: Principal Investigator, Jingyun Wang, Assistant Professor, Salus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HJW1602
Record Dates: First submitted 2016-02-16; First posted 2016-02-22 (Estimated); Results first posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia | interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12-hour IO-therapy Glasses (Experimental): wear IO-therapy glasses for 12-hour
  Interventions: Device: IO-therapy Glasses
- 6-hour patching (Active Comparator): wear the eye patch for 6-hour
  Interventions: Device: patch

INTERVENTIONS:
Device: IO-therapy Glasses — 12-hour of 50% intermittent occlusion therapy on the fellow eye.
  Arms: 12-hour IO-therapy Glasses
Device: patch — 6-hour of eye patch on the fellow eye
  Arms: 6-hour patching

SUMMARY:
This study is designed to evaluate the effectiveness of a novel amblyopia treatment - Intermittent occlusion therapy (IO-therapy) glasses (AmblyzTM) in treating severe amblyopia.

Children ages 3 to 8 years with severe amblyopia (visual acuity of 20/100 to 20/400 in the amblyopic eye) will be enrolled and randomized into two groups: 1) standard 6-hour patching group or 2) 12-hour IO-therapy glasses group.

The study also observe the effectiveness of IO-therapy glasses on two types of difficult amblyopia: deprivation amblyopia associated with congenital or developmental cataract, and myopic anisometropic amblyopia.

DETAILED DESCRIPTION:
Children ages 3 to < 8 years with severe/dense amblyopia (visual acuity of 20/100 to 20/400 in the amblyopic eye) will be enrolled and randomized into two groups: 1) standard 6-hour patching group or 2) 12-hour IO-therapy glasses group.

Children ages 3 to < 8 years with deprivation amblyopia associated with congenital or developmental cataracts (visual acuity of 20/40 to 20/400 in the amblyopic eye) will be enrolled.

Children ages 3 to < 8 years with myopic anisometropic amblyopia will be enrolled into an intermittent occlusion therapy glasses (AmblyzTM) group.

According to visual acuity, they will receive one of two IO-therapy glasses treatment regimens: 1) If the amblyopic eye is between 20/40 to 20/80 inclusive, 4-hour IO-therapy glasses or 2) If the amblyopic eye is between 20/100 to 20/400 inclusive, the child will receive12-hour IO-therapy glasses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 to < 8 years
2. Amblyopia associated with strabismus, anisometropia, or both
3. Visual acuity, measured in each eye without cycloplegia within 7 days prior to enrollment using the ATS single-surround HOTV letter protocol as follows:

   * Visual acuity in the amblyopic eye between 20/100 and 20/400 inclusive
   * Visual acuity in the sound eye 20/32 or better
4. Spectacle correction (if applicable) for measurement of enrollment visual acuity must meet the following criteria and be based on a cycloplegic refraction within 6 months:

   * Requirements for spectacle correction:
   * For patients meeting criteria for only strabismus i. Hypermetropia if corrected must not be undercorrected by more than +1.50 D spherical equivalent, and the reduction in plus sphere must be symmetric in the two eyes. Otherwise, spectacle correction is at investigator discretion.
   * For patients meeting criteria for anisometropia or combined-mechanism i. Spherical equivalent must be within 0.50 D of fully correcting the anisometropia ii. Hypermetropia must not be undercorrected by more than +1.50 D spherical equivalent, and reduction in plus must be symmetric in the two eyes iii. Cylinder power in both eyes must be within 0.50 D of fully correcting the astigmatism iv. Cylinder axis in the spectacle lenses in both eyes must be within 6 degrees of the axis of the cycloplegic refraction
5. Wearing optimal spectacle correction for a minimum of 4 weeks at the time of enrollment.
6. Gestational age > 34 weeks and birth weight > 1500 grams
7. Parent willing to accept randomization
8. Parent willing to be contacted and has access to phone
9. Parent does not anticipate relocation outside area of active study site

Exclusion Criteria:

* • Amblyopic eye has myopia worse than -3.00D spherical equivalent.

  * Previous amblyopia treatment within 6 months.
  * Prior intraocular or refractive surgery
  * Known skin reactions to patch or bandage adhesives
  * Systemic diseases that may cause reduced vision such as Down syndrome.

If patients are in the deprivation amblyopia category, the following criteria must be met for the patient to be enrolled in the study:

1. Age 3 to < 8 years
2. Amblyopia due to previous congenital or developmental cataract surgery.
3. Visual acuity, measured in each eye without cycloplegia within 7 days prior to enrollment using the ATS single-surround HOTV letter protocol as follows:

a. Visual acuity in the amblyopic eye between 20/40 and 20/400 inclusive b. Visual acuity in the sound eye 20/32 or better c. Inter-eye acuity difference ≥ 2 logMAR lines (i.e., amblyopic eye acuity at least 3 lines worse than sound eye acuity) d) Gestational age > 34 weeks and birth weight > 1500 grams e) Parent willing to be contacted and has access to phone.

If patients are enrolled in the myopic anisometropia amblyopia category, the following criteria must be met for the patients to be enrolled in the study.

* Aged 3 to <8 years
* Best-corrected VA in the amblyopic eye of 20/40 to 20/400 inclusive
* Best-corrected VA in the fellow eye of 20/40 or better
* Magnitude of myopic anisometropia of > 3.00 D
* Intereye acuity difference of > 3 logMAR lines
* Amblyopia associated with myopic anisometropia
* Has been wearing optimal spectacle correction for a minimum of four weeks

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jingyun Wang, PhD, Principal Investigator — Salus University
Locations (1):
- Salus University, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Deprivation Amblyopia: This group observes if the patients with deprivation amblyopia (amblyopia post-cataract surgery) could improve with IO-therapy glasses.
- Myopic Anisometropic Amblyopia: This group observes if patients with myopic anisometropic amblyopia can improve vision with IO-therapy glasses
Period: Overall Study
Arm/Group | 12-hour IO-therapy Glasses | 6-hour Patching | Deprivation Amblyopia | Myopic Anisometropic Amblyopia
Started | 6 | 6 | 2 | 4
Completed | 2 | 4 | 2 | 3
Not Completed | 4 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0
Not completed — the device is too small for the patient. | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Deprivation Amblyopia; Myopic Anisometropic Amblyopia: wear IO-therapy glasses depends on the severity of amblyopia. If severe, wear 12 hours; if moderate, wear 4 hours.
- Total: Total of all reporting groups
Arm/Group | 12-hour IO-therapy Glasses | 6-hour Patching | Deprivation Amblyopia | Myopic Anisometropic Amblyopia | Total
Number analyzed (Participants) | 2 | 4 | 2 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: Year] | 4.7 (0.2) | 5.4 (1.6) | 6.8 (0.1) | 5.9 (0.6) | 5.7 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 2 | 6
  Male | 1 | 2 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 2 | 3 | 1 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 3 | 3
  White | 2 | 4 | 2 | 0 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
visual acuity of amblyopic eye [Mean (Standard Deviation); unit: logMAR] — visual acuity was measured with ATS-HOTV methods. it is described with logMAR value. The higher value is, the worse the vision of the eye is.
  logMAR | 1.10 (0.28) | 0.86 (0.17) | 0.75 (0.35) | 0.5 (0.17) | 0.71 (0.29)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Improvement
Description: Visual acuity was measured with ATS-HOTV methods in logMAR. The larger amount means the worse acuity. Visual acuity improvement is defined as the change at the primary outcome follow-up visit from the baseline. (Note: Visual acuity improvement = Visual acuity at the baseline - Visual acuity at the 12-week follow-up) The larger amount of change indicates better improvement.
Time Frame: 12± 1 weeks after treatment
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Deprivation Amblyopia: This group observes the efficacy of IO-therapy glasses in children with deprivation amblyopia (amblyopia post-cataract surgery).
- Myopic Anisometropic Amblyopia: This group observes the efficacy of IO-therapy glasses in children with myopic anisometropic amblyopia.
Arm/Group | 12-hour IO-therapy Glasses | 6-hour Patching | Deprivation Amblyopia | Myopic Anisometropic Amblyopia
Number analyzed (Participants) | 2 | 4 | 2 | 3
logMAR | 0.05 (0.07) | 0.17 (0.23) | 0.05 (0.07) | 0.1 (0.26)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: reverse amblyopia Reverse amblyopia is defined as, at the follow-up visit, the good fellow eye's visual acuity being two logMAR lines worse than the baseline.
Arm/Group | 12-hour IO-therapy Glasses | 6-hour Patching | Deprivation Amblyopia | Myopic Anisometropic Amblyopia
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/3

LIMITATIONS AND CAVEATS:
This trial is limited in enrollment. The device has only one size and it did not fit a patient in the Amblyz group. We are not sure if some patients in that group lost follow-up because of the size of the glasses.

Due to the small sample size, we are not able to draw a conclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT02687581/Prot_SAP_ICF_000.pdf